CLINICAL TRIAL: NCT02931851
Title: Family Information Management in the Intensive Care Unit: A Randomized Controlled Trial
Brief Title: Family Information Management in the Intensive Care Unit
Acronym: ICU-Families
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Medical University of Vienna (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ICU-Families 1.0
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Extended Family

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Standard Information
  Interventions: Other: Placebo
- Intervention (Active Comparator): Professionally developed website for relatives of ICU patients
  Interventions: Other: ICU Families Website

INTERVENTIONS:
Other: ICU Families Website — Professionally developed website for relatives of ICU patients
  Arms: Intervention
Other: Placebo — Standard Information provided online
  Arms: Placebo

SUMMARY:
Relatives in intensive care units (ICU) are important partners in decision-making in the treatment of critically ill patients and provide a significant resource in the care and recovery of patients. Therefore, a professional, educational intervention targeting these caregivers may have fundamental benefits with little risk. As in other fields, information is searched in the internet, but this unselected information is often overwhelming and of little use in this context.

Symptoms of anxiety, stress and depression are common in affected relatives. The majority of family members report some level of anxiety, depression and stress, sometimes even resulting in post-traumatic stress disorder (PTSD). Importantly, an association between lack of information and post-traumatic stress disorder PTSD has been reported. The large number of potentially affected families poses a particular challenge to healthcare and may cause substantial secondary costs to national economy.

DETAILED DESCRIPTION:
Design:

1. Phase: Empirical study (quantitative) of information needs - semi-structured interviews with family members, physicians and caregivers
2. Phase: Development of user friendly homepage with University of Applied Sciences Joanneum and validation of the homepage with medical professionals and laypersons
3. Phase: Randomized Controlled Trial (non-blinded) with "placebo home page" (N=110)

Background:

Relatives in intensive care units (ICU) are important partners in decision-making in the treatment of critically ill patients and provide a significant resource in the care and recovery of patients. Therefore, a professional, educational intervention targeting these caregivers may have fundamental benefits with little to no risk. As in other fields, information is searched in the internet, but this unselected information is often overwhelming and of little use in this context.

In Austria there are 2784 systemized intensive care beds with an average occupation of 3,6 days, representing 100 new admissions per year/ICU bed. This may translate to 500.000 affected family members per year.

The role of family members in the treatment process of ICU patients is a not very well studied subject, especially in German-speaking countries. In contrast, in the Anglo-American world, family members play a key role in the medical, financial and legal aspects of the treatment process and have a decisive role in the successful treatment during and after critical illness.

Symptoms of anxiety, stress and depression are common in affected relatives . The majority of family members report some level of anxiety, depression and stress, sometimes even resulting in post-traumatic stress disorder (PTSD). Importantly, an association between lack of information and post-traumatic stress disorder PTSD has been reported. The large number of potentially affected families poses a particular challenge to healthcare and may cause substantial secondary costs to national economy.

The participation of relatives in the decision making process of ICU patients is negatively affected by the uncertainty concerning the treatment path, medical procedures and consequences for the families' life after ICU discharge. This likely leads to unnecessary hospital readmissions, complicates rehabilitation of patients and requires adapted management strategies for relatives. Therefore, it is important to provide sufficient information to families in high quality.

The relationship management with relatives places significant demands on ICU staff and conflicts between physicians and relatives are common. So far, only a few randomized intervention studies have been performed in this setting, but with promising results.

The internet has revolutionized our world including the access to medical information. In one study, almost 50% of ICU patients' family members used the internet for information purposes within the first days of ICU treatment. This makes a web-based intervention in this setting very promising. To our knowledge however, no RCT has yet evaluated the usefulness of a web-based intervention on ICU patients' family members' quality of life.

The following question should therefore be answered by our study:

* Does targeted information and communication using new media (INTERVENTION) have a beneficial influence on subjective and objective endpoints of patients and their families?
* Could this help in averting the negative effects of anxiety, stress, and depression? Are new media accepted in clinical routine?
* Does the project support the affected family members in their health literacy?

ELIGIBILITY:
Inclusion Criteria:

* anticipated further ICU stay ≥3 days (index patient)

Exclusion Criteria:

* lack of Basic Information Technology (IT) user knowledge or German language skills
* DNR (Do not resuscitate) orders (index patient)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Subjective distress | 30 Days
  Impact of Event Score (IES: symptoms of post traumatic stress disorder)

SECONDARY OUTCOMES:
Levels of anxiety and depression | 30 days
  Measured by Hospital Anxiety and Depression Score (HADS)
Subjective usefulness of the website for relatives | 30 days
  Subjective Evaluation
Length of stay | 90 days
  ICU and Hospital length of stay of the index patients
Readmissions | 90 days
  number of readmissions of the index patients
Mortality | 90 days
  mortality of the index patients
User-statistics | 30 days
  user statistics for the website

CONTACTS AND LOCATIONS:
Overall Officials: Karin Amrein, MD, MSc, Principal Investigator — Medical University of Graz
Locations (3):
- Austria (2):
  - Medical University of Graz, Graz
  - Medical University of Vienna, Vienna
- University of Berne - Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Azoulay E, Kentish-Barnes N, Nelson JE. Communication With Family Caregivers in the Intensive Care Unit: Answers and Questions. JAMA. 2016 May 17;315(19):2075-7. doi: 10.1001/jama.2016.5637. No abstract available. PMID 27187298
- [Background] Peigne V, Chaize M, Falissard B, Kentish-Barnes N, Rusinova K, Megarbane B, Bele N, Cariou A, Fieux F, Garrouste-Orgeas M, Georges H, Jourdain M, Kouatchet A, Lautrette A, Legriel S, Regnier B, Renault A, Thirion M, Timsit JF, Toledano D, Chevret S, Pochard F, Schlemmer B, Azoulay E. Important questions asked by family members of intensive care unit patients. Crit Care Med. 2011 Jun;39(6):1365-71. doi: 10.1097/CCM.0b013e3182120b68. PMID 21358395
- [Background] Lautrette A, Darmon M, Megarbane B, Joly LM, Chevret S, Adrie C, Barnoud D, Bleichner G, Bruel C, Choukroun G, Curtis JR, Fieux F, Galliot R, Garrouste-Orgeas M, Georges H, Goldgran-Toledano D, Jourdain M, Loubert G, Reignier J, Saidi F, Souweine B, Vincent F, Barnes NK, Pochard F, Schlemmer B, Azoulay E. A communication strategy and brochure for relatives of patients dying in the ICU. N Engl J Med. 2007 Feb 1;356(5):469-78. doi: 10.1056/NEJMoa063446. PMID 17267907
- [Derived] Hoffmann M, Jeitziner MM, Riedl R, Mueller G, Peer A, Bachlechner A, Heindl P, Burgsteiner H, Schefold JC, von Lewinski D, Eller P, Pieber T, Sendlhofer G, Amrein K. Effects of an online information tool on post-traumatic stress disorder in relatives of intensive care unit patients: a multicenter double-blind, randomized, placebo-controlled trial (ICU-Families-Study). Intensive Care Med. 2023 Nov;49(11):1317-1326. doi: 10.1007/s00134-023-07215-4. Epub 2023 Oct 23. PMID 37870597